CLINICAL TRIAL: NCT02740010
Title: Retrospective Observational Trial on the Visual Performances of a Progressive Multifocal Intraocular Lens With Extended Depth of Focus
Brief Title: The Visual Performances of a Progressive Multifocal Intraocular Lens With Extended Depth of Focus
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: PSM8
Record Dates: First submitted 2016-04-04; First posted 2016-04-15 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cataract; Presbyopia
Keywords: extended depth of focus; cataract surgery; presbyopia correction
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: EDOF Mini WELL Ready IOL — implant

SUMMARY:
The purpose of this observational, non-controlled, multicenter trial with a retrospective design is to evaluate the visual performance of one cohort of patients who received the EDOF MINI WELL® intraocular lenses following refractive lens exchange (RLE) or cataract surgery.

DETAILED DESCRIPTION:
The study aims at evaluating the visual performance of the EDOF MINI WELL® in qualitative and quantitative terms of the progressive vision. The cohort of subjects includes all patients submitted in the six involved Centers. for the surgical procedure for cataract extraction or Refractive Lens Exchange (RLE) using the MINI WELL® with a pre-operative visit (from the day - 60 to day -1 before surgery) and a post-operative follow-up visit performed 30-60 days after implant.

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age above 18 years
* Refractive lens exchange (RLE) or cataract surgery
* Symmetrical preoperative keratometric astigmatism < 0.75 D
* Healthy corneas, not treated surgically

Exclusion Criteria:

* Previous corneal surgery (i.e. pterygium, refractive surgery)
* Eye diseases with visual acuity < 20/32
* Pseudoexfoliation
* Abnormal pupil size and position.
* Use of contact lens 30 days before the preoperative visit.
* Corneal warpage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone cataract or RLE surgery with the IOL MINI WELL and having a post-operative follow up visit (30-60 days) in the period from March, 1st 2014 to March,31st 2016.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Refraction; UDVA (Uncorrected Distance Visual Acuity); CDVA (Corrected Distance Visual Acuity); DCNVA (Distance Corrected Near Visual Acuity); Defocus curve; Reading speed; Halometry. | 60 days

SECONDARY OUTCOMES:
Adverse Device Effects (ADE); Serious Adverse Device Effects (SADE); Unexpected Serious Adverse Device Effects (USADE); Adverse Events (AE); Serious Adverse Events (SAE). | 60 days

OTHER OUTCOMES:
Contrast sensitivity | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dominguez-Vicent A, Esteve-Taboada JJ, Del Aguila-Carrasco AJ, Ferrer-Blasco T, Montes-Mico R. In vitro optical quality comparison between the Mini WELL Ready progressive multifocal and the TECNIS Symfony. Graefes Arch Clin Exp Ophthalmol. 2016 Jul;254(7):1387-97. doi: 10.1007/s00417-015-3240-7. Epub 2015 Dec 16. PMID 26671689
- [Background] Dominguez-Vicent A, Esteve-Taboada JJ, Del Aguila-Carrasco AJ, Monsalvez-Romin D, Montes-Mico R. In vitro optical quality comparison of 2 trifocal intraocular lenses and 1 progressive multifocal intraocular lens. J Cataract Refract Surg. 2016 Jan;42(1):138-47. doi: 10.1016/j.jcrs.2015.06.040. PMID 26948789
- [Background] Packer M, Fine IH, Hoffman RS. Aspheric intraocular lens selection: the evolution of refractive cataract surgery. Curr Opin Ophthalmol. 2008 Jan;19(1):1-4. doi: 10.1097/ICU.0b013e3282f2d791. No abstract available. PMID 18090888
- [Background] Kohnen T, Klaproth OK, Buhren J. Effect of intraocular lens asphericity on quality of vision after cataract removal: an intraindividual comparison. Ophthalmology. 2009 Sep;116(9):1697-706. doi: 10.1016/j.ophtha.2009.03.052. Epub 2009 Jul 29. PMID 19643497
- [Background] Lehmann R, Waycaster C, Hileman K. A comparison of patient-reported outcomes from an apodized diffractive intraocular lens and a conventional monofocal intraocular lens. Curr Med Res Opin. 2006 Dec;22(12):2591-602. doi: 10.1185/030079906X158039. PMID 17166341
- [Background] Leyland M, Zinicola E. Multifocal versus monofocal intraocular lenses in cataract surgery: a systematic review. Ophthalmology. 2003 Sep;110(9):1789-98. doi: 10.1016/S0161-6420(03)00722-X. PMID 13129879
- [Background] Steinert RF. Visual outcomes with multifocal intraocular lenses. Curr Opin Ophthalmol. 2000 Feb;11(1):12-21. doi: 10.1097/00055735-200002000-00004. PMID 10724823
- [Background] Blaylock JF, Si Z, Vickers C. Visual and refractive status at different focal distances after implantation of the ReSTOR multifocal intraocular lens. J Cataract Refract Surg. 2006 Sep;32(9):1464-73. doi: 10.1016/j.jcrs.2006.04.011. PMID 16931257
- [Background] Maxwell WA, Cionni RJ, Lehmann RP, Modi SS. Functional outcomes after bilateral implantation of apodized diffractive aspheric acrylic intraocular lenses with a +3.0 or +4.0 diopter addition power Randomized multicenter clinical study. J Cataract Refract Surg. 2009 Dec;35(12):2054-61. doi: 10.1016/j.jcrs.2009.06.041. PMID 19969208
- [Background] Munoz G, Albarran-Diego C, Ferrer-Blasco T, Sakla HF, Garcia-Lazaro S. Visual function after bilateral implantation of a new zonal refractive aspheric multifocal intraocular lens. J Cataract Refract Surg. 2011 Nov;37(11):2043-52. doi: 10.1016/j.jcrs.2011.05.045. PMID 22018366
- [Background] Pepose JS, Qazi MA, Chu R, Stahl J. A prospective randomized clinical evaluation of 3 presbyopia-correcting intraocular lenses after cataract extraction. Am J Ophthalmol. 2014 Sep;158(3):436-46.e1. doi: 10.1016/j.ajo.2014.06.003. Epub 2014 Jun 14. PMID 24932989
- [Background] Jiang T, Jiang J, Zhou Y, Zhao GQ, Li H, Zhao SY. Cataract surgery in aged patients: phacoemulsification or small-incision extracapsular cataract surgery. Int J Ophthalmol. 2011;4(5):513-8. doi: 10.3980/j.issn.2222-3959.2011.05.11. Epub 2011 Oct 18. PMID 22553713